CLINICAL TRIAL: NCT00674310
Title: A Single-Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Ropinirole 0.25 mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Richard Larouche, M.D., SFB C Anapharm
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROPI-T25-PVFD-1
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease; Restless Leg Syndrome
MeSH Terms: conditions — Parkinson Disease; Restless Legs Syndrome | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole Hydrochloride — Restless Leg Syndrome

SUMMARY:
The objective of this study was to assess the single dose bioequivalence of Roxane's Ropinirole tablets,0.25 mg, to ReQuip Tablets, 0.25 mg (GlaxoSmithKline) under fed conditions using a single dose, randomized, 2-treatment, 2-period, 2-sequence cross-over design.

DETAILED DESCRIPTION:
The objective of this study was to assess the single dose bioequivalence of Roxane's Ropinirole tablets,0.25 mg, to ReQuip Tablets, 0.25 mg (GlaxoSmithKline) under fed conditions using a single dose, randomized, 2-treatment, 2-period, 2-sequence cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to ropinirole or any other comparable product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2004-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, M.D., Principal Investigator — SFBC Anapharm